CLINICAL TRIAL: NCT01437943
Title: P-MR Spectroscopy Evaluation of the Effect of Short-Term Treatment With Aliskiren on Kidney β-ATP/Pi Level in Kidney Transplant Patients
Brief Title: Effect of Short Term Aliskiren Treatment in Kidney Transplant Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Novartis has have decided to terminate all clinical investigator-initiated research projects involving aliskiren
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Anil K. Chandraker, MD, Medical Director of Renal Transplantation, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010P000005
Record Dates: First submitted 2011-09-20; First posted 2011-09-21 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-03

CONDITIONS: Kidney Disease; Kidney Failure, Chronic
Keywords: Transplant; Failure; Kidney
MeSH Terms: conditions — Kidney Diseases; Kidney Failure, Chronic | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren (Active Comparator): Aliskiren 150 mg daily for 180 days
  Interventions: Drug: Aliskiren
- Placebo (Placebo Comparator): Placebo identical to Aliskiren drug daily for 180 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aliskiren — Take 1 tablet (150 mg) by mouth daily for 180 days
  Other Names: Tekturna
  Arms: Aliskiren
Drug: Placebo — Take 1 tablet (0 mg) daily for 180 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of a short-term aliskiren treatment on kidney metabolism in patients at high risk for developing kidney dysfunction (i.e. kidney transplanted patients). The study is aimed at evaluating if any effect on kidney metabolism [using proton MR Spectroscopy(1H-MRS)] can be detected following a 6 months treatment with aliskiren regardless of its anti-hypertensive role. 1H-MRS can record a larger number of chemical species (up to 40) in the kidney, and monitor changes according to the pathologic state and health of the transplanted kidney.

ELIGIBILITY:
Inclusion Criteria:

* Stable patients with end stage renal disease receiving cadaveric kidney transplantation will be enrolled. Patients must have at least 6 months of follow-up to be included in the study. Patients must have stable creatinine levels in the last 6 months (no change>0.5 mg/dl).
* Patients with a systolic blood pressure of 120 or above

Exclusion Criteria:

* Serum potassium > 5.0 mmol/L (at the visit directly preceding Randomization);
* History of any cardiovascular event (stroke, TIA, MI, unstable angina, CABG, percutaneous coronary intervention, hospitalization due to HF) during the 3 months prior to Visit 1. If a patient experiences such an event between Visit 1 and randomization at Visit 3, he/she should be withdrawn from the screening phase. If suitable, the patient can be re-screened at a later stage;
* Hypertension (at enrollment): any patient with msSBP ≥ 170 mmHg or msDBP ≥ 110 mmHg;
* Congestive heart failure NYHA class III and IV;
* Concomitant treatment with two (2) or more renin-angiotensin-aldosterone system blocking agents, e.g. ACEI, ARB or aldosterone-antagonist;
* Unstable serum creatinine, no patients with creatinine >2.5 mg/dl will be enrolled;
* Second (II) or third (III) degree heart block without a pacemaker;
* Concurrent potentially life threatening arrhythmia or other uncontrolled arrhythmia;
* Clinically significant valvular heart disease;
* Known renal artery stenosis;
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of the study drugs including, but not limited to, any of the following: (i) History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection (patients with previous bariatric surgery > 6 months prior to Visit 1 are allowed to participate); (ii) Any history of pancreatic injury, pancreatitis or evidence of impaired pancreatic function/injury as indicated by abnormal lipase or amylase; (iii) Evidence of hepatic disease as determined by any one of the following: SGPT value exceeding 3 x Upper Limit of Normal (ULN) at Visit 1, a history of hepatic encephalopathy, a history of cirrhosis, esophageal varices, or a history of portocaval shunt.
* History of malignancy other than basal cell skin cancer within the past five years.
* Any concurrent life threatening condition with a life expectancy less than 2 years.
* History or evidence of drug or alcohol abuse within the last 12 months.
* Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.
* History of hypersensitivity to any of the study drugs or to medications belonging to the same therapeutic class as the study drugs as well as known or suspected contraindications to the study drugs.
* History of noncompliance to medical regimens or unwillingness to comply with the study protocol.
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer
* Any condition that in the opinion of the investigator would jeopardize the evaluation of efficacy or safety.
* Persons directly involved in the execution of this protocol.
* Pregnant or nursing (lactating) women
* Women of Child-Bearing Potential (WOCBP) unless postmenopausal for at least one year, surgically sterile or using effective methods of contraception as defined by local Health Authorities.
* Treatment with Cyclosporine.

Exclusion criteria include MR contraindications:

* electrical implants such as cardiac pacemakers or perfusion pumps
* ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants
* ferromagnetic objects such as jewelry or metal clips in clothing
* pregnant volunteers
* pre-existing medical conditions including a likelihood of developing seizures or claustrophobic reactions
* any greater than normal potential for cardiac arrest
* subjects less than 18 years of age.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anil Chandraker, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 subjects were recruited into the trial however none completed the treatment/follow-up as Novartis terminated all studies involving Aliskiren.
Groups:
- Placebo: Placebo daily for 180 days
  Placebo: Take 1 tablet by mouth daily for 180 days
Period: Overall Study
Arm/Group | Aliskiren | Placebo
Started | 7 | 3
Completed | 0 | 1
Not Completed | 7 | 2
Not completed — Aliskiren trials terminated by Novartis | 4 | 2
Not completed — Subject expressed pregnancy plans | 1 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo daily for 180 days
  Placebo: Take 1 tablet (0 mg) daily for 180 days
- Total: Total of all reporting groups
Arm/Group | Aliskiren | Placebo | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 56.6 [42 to 75] | 48 [33 to 64] | 54 [33 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 6 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Effect of Aliskiren on Kidney Metabolism
Description: Evaluation of aliskiren on kidney metabolism by P-MR spectroscopy
Time Frame: 180 days (completion of treatment)
Population: Only one subject completed study drug and no subjects had completed the 6 month P-MR scan at the time the trial was terminated. Because of this, we were not able to analyze the primary outcome.
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected continuously during subject participation starting at consent through month 6 or termination of the trial.
Arm/Group | Aliskiren | Placebo
Serious Adverse Events (participants affected / at risk) | 2/7 | 1/3
Other Adverse Events (participants affected / at risk) | 5/7 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aliskiren (N=7) | Placebo (N=3)
GI bleed (Gastrointestinal disorders) | 1 (2) | 0 (0) — possible diverticulitis
Left knee hemarthrosis and DVT (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — s/p left knee arthroscopy
Salmonella group B (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren (N=7) | Placebo (N=3)
Diarrhea (Gastrointestinal disorders) | 5 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Urinary tract infection (Renal and urinary disorders) | 0 | 1
Hypotension (Cardiac disorders) | 0 | 1
Lower extremity weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Elevated creatinine (Renal and urinary disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
In December 2011, all studies involving Aliskiren were terminated by Novartis after interim analysis of the ALTITUDE trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No